CLINICAL TRIAL: NCT05311527
Title: Using UroLift System With Stereotactic Ablative Body Radiotherapy For Men With Prostate Cancer and Benign Prostatic Hyperplasia (BPH): a Phase I Safety Trial
Brief Title: UroLift System With SAbR for Prostate Cancer and BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: NeoTract, Inc. (Industry)
Responsible Party: Principal Investigator, Aurelie Garant, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0261
Record Dates: First submitted 2022-03-15; First posted 2022-04-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Masking Description: Non-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All Study participants (Experimental): Study participants will undergo Urolift System followed by SABR
  Interventions: Device: Urolift; Radiation: SABR

INTERVENTIONS:
Device: Urolift — Urolift Implant
Radiation: SABR — Stereotactic Body Radiation Therapy for prostate cancer
  Other Names: SBRT

SUMMARY:
Confirming safety of combining UroLift System prior to SAbR for patients with newly diagnosed prostate cancer and a history of BPH, by measuring the acute complication rate of UroLift System implant in patients with BPH undergoing SAbR (within 90 days of treatment completion)

DETAILED DESCRIPTION:
UroLift System implant will be implanted transurethrally under cystoscopic guidance with a UroLift System Delivery Device by a trained provider. Optimal placement of the implants will be verified cystoscopically. On average, 4-6 UroLift System implants are typically implanted but more or less can be placed per provided discretion, up to a maximum of 10 implants per manufacturer specifications.

Given that patients will also undergo UroLift System placement, patients will be offered to undergo UroLift System, fiducial marker placement and rectal gel spacer placement in one single procedure, under general anesthesia.

SAbR will be performed following placement of UroLift System, prostate fiducials, rectal spacer, and MR/CT simulation, using stereotactic immobilization/localization, rectal enema, prophylactic medication support (tamsulosin, dexamethasone unless contraindicated), bladder filling protocol, and appropriate imaging verification.

ELIGIBILITY:
Inclusion Criteria:

* AJCC 8th edition clinical stage T1 (a, b, or c) or T2 (a, b, or c) adenocarcinoma of the prostate gland, Gleason 3+3 = 6 or 3+4 = 7, with no direct evidence of regional or distant metastases following appropriate staging studies. See Appendix I for details on AJCC 8th Edition staging criteria. T-staging may be assessed by multi-parametric imaging alone if digital rectal examination was deferred
* Histologic confirmation of prostate cancer is required by biopsy performed within 18 months of registration.
* Age ≥ 45 years.
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-1.
* American Society of Anesthesia (ASA) physical status score of 1-3
* Baseline AUA symptom score ≥ 17 regardless of medical therapy
* The serum PSA should be ≤ 20 ng/ml within 120 days of registration
* Study entry PSA must not be obtained during the following time frames: (1) 10-day period following prostate biopsy; (2) following initiation of ADT or anti-androgen therapy; (3) within 30 days after discontinuation of finasteride; (4) within 90 days after discontinuation of dutasteride; (5) within 5 days of a digital rectal examination
* Ultrasound or MRI based volume estimation of prostate gland < 100 grams, regardless of cytoreduction with pharmacotherapy
* Ability to undergo general anesthesia for <60 minutes
* Ability to understand and the willingness to sign a written informed consent.
* All men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

Exclusion Criteria:

* Contraindications to UroLift System placement including:
* Prostate volume >100 cc based on imaging-based estimation
* Urethral conditions (e.g. urethral strictures and neoplams) that may prevent insertion of UroLift System delivery system into the bladder
* Urinary incontinence due to incompetent sphincter
* An active urinary tract infection
* Current gross hematuria

In addition to the contraindications if there is a known allergy to nickel, titanium, or stainless steel these patients should be excluded

* Prior transurethral resection of the prostate (TURP), median lobe manipulation, simple prostatectomy, or other ablative procedures for benign prostatic hyperplasia.
* Foley / self-catheterization in the last 12 months.
* Patients with all three intermediate risk factors (PSA >10 and ≤ 20, Gleason 7, clinical stage T2b-T2c) who ALSO have ≥50% of the number of their template biopsy cores positive for cancer are ineligible.
* Prior pelvic radiotherapy, chemotherapy, or surgery for prostate cancer.
* Current active androgen deprivation therapy

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Safety of UroLift implant when combined with SAbR for men with prostate cancer and benign prostatic hyperplasia | 90 days
  Analyses will be performed for all subjects having received at least one fraction of radiation therapy. The study will use CTCAE version 5.0 for reporting of adverse events and, for reporting purposes, will also capture Clavien-Dindo grading system for the classification of surgical complications for reporting adverse events related to the UroLift System procedure.

SECONDARY OUTCOMES:
Quality of Life with UroLift System | 90 days
  AUA, EPIC-26 questionnaires and Noninvasive urodynamics will be obtained, these data will be analyzed once all patients have completed the scheduled trial visits.The aggregate score will be done for (urinary, sexual, bowel, and health-related) associated with UroLift System when administered prior to SABR.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie Garant, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States